CLINICAL TRIAL: NCT04271683
Title: Safe Use of CPAP During Preoxygenation and PEEP After Apnoea During Induction of General Anesthesia
Brief Title: Safe Use of CPAP and PEEP During Induction of General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Lennart Edmark, Consultant, Principal Investigator, Region Västmanland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPM 2019-05092
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: General Anesthesia
Keywords: Positive end-expiratory pressure; Mechanical ventilation; Induction of anesthesia
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure controlled ventilation with PEEP (Experimental): In this group, ventilation after apnoea during induction of general anesthesia starts with pressure controlled ventilation with PEEP.
  Interventions: Procedure: Pressure controlled ventilation with PEEP
- Manual ventilation without PEEP (Active Comparator): In this group, ventilation after apnoea during induction of general anesthesia starts with manual ventilation without PEEP.
  Interventions: Procedure: Manual ventilation without PEEP

INTERVENTIONS:
Procedure: Pressure controlled ventilation with PEEP — The intervention consists of starting ventilation after apnoea during induction of general anesthesia with pressure controlled ventilation with PEEP instead of manually without PEEP.
  Arms: Pressure controlled ventilation with PEEP
Procedure: Manual ventilation without PEEP — The intervention consists of starting ventilation after apnoea during induction of general anesthesia manually instead of with pressure controlled ventilation with PEEP.
  Arms: Manual ventilation without PEEP

SUMMARY:
The study compares the safety of using pressure controlled ventilation with a positive end-expiratory pressure (PEEP) during induction of general anaesthesia immediately after apnoea to a standard method starting ventilation manually without PEEP immediately after apnoea.

DETAILED DESCRIPTION:
Using a continuous positive pressure (CPAP) during preoxygenation, followed by pressure controlled ventilation with PEEP after apnoea during induction of general anesthesia, might offer several benefits but safety issues needs more investigation. This study compares the safety of using pressure controlled with PEEP during induction of general anesthesia immediately after apnoea to a standard method starting ventilation manually without PEEP immediately after apnoea.

ELIGIBILITY:
Inclusion Criteria:

* Normal or overweight patients scheduled for day case surgery in general anesthesia.
* American Society of Anesthesiologists functional class I-III.
* Body Mass Index 18.5-30.

Exclusion Criteria:

* Increased risk of regurgitation of gastric content.
* Symptomatic asthma, COPD or heart failure.
* Peripheral oxygen saturation (SpO2) breathing air <94 %
* Anticipated difficult airway.
* Beard.
* Anatomical features making it difficult to keep a tight seal during maskventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Number of breaths until return of CO2. | 2 minutes
  When starting ventilation after apnea the number of breaths given until the return of CO2 is at least 1.3 kPa at a respiratory frequency of 10 per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Edmark, PhD, Principal Investigator — Region Västmanland
Locations (1):
- Lennart Edmark, Västerås, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Please email request to the study principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after publication of study results, approximately 18 months after study completion.
Access Criteria: Data access requests will be reviewed by a review panel at the Center for Clinical Research, Västerås.
  Requestors will be required to sign a data access agreement.
  .